CLINICAL TRIAL: NCT06842004
Title: Protocol to Improve the Representation of the Reproductive Process in Spanish Fiction: Sequential Transformative Approach, With Qualitative Predominance and Participatory Action.
Brief Title: Protocol to Improve the Representation of the Reproductive Process in Spanish Fiction.
Acronym: MaterScreen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Rosa Mar Alzuria Alós, Rn, RM, PhD, Universitat de Lleida
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PID2022-137338OA-I00; PID2022-137338OA-I00 (Other Grant/Funding Number: Ministerio de Ciencia e Innovación, Gobierno de España)
Record Dates: First submitted 2025-01-31; First posted 2025-02-24 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Sexual Health; Community Participation; Social Norms
Keywords: sexual health; motion pictures; community participation; social norms

STUDY DESIGN:
Intervention Model Description: The study will employ a sequential mixed-methods transformative design (DITRAS), with a predominantly qualitative approach and a strong emphasis on participatory action research. It will be structured into three distinct phases.
  In the first phase, a quantitative approach will be used, involving a descriptive cross-sectional study based on a systematic search of film databases, digital platforms, and on-demand television.
  The second phase will focus on exploring the perceptions of users and professionals regarding reproductive health processes through focus groups and interviews.
  The third phase, the intervention phase, will adopt a participatory action research approach to co-create a good practice manual, which will be implemented in undergraduate and postgraduate communication and journalism training programs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Persons involved in reproductive processes (Other): The participatory action in this mixed study will be applied to users, health professionals and audiovisual professionals to co-create solutions and reflect on the representations of motherhood in Spanish audiovisual fiction. This methodology seeks to actively involve those involved-health professionals, audiovisual experts and people with experience in maternity-in all phases of the study, from data collection to interpretation.
  Interventions: Other: Participatory action

INTERVENTIONS:
Other: Participatory action — The reality of audiovisual fiction in Spain and professionals' perceptions of how motherhood is portrayed will be explored. Through participatory action, participants will share their experiences and knowledge to identify areas for improvement in the representation of reproductive processes. The result will be a manual of good practices for fiction production, aimed at promoting more inclusive, realistic and stereotype-free representations, in order to improve both public perception and professional training in the audiovisual field.

SUMMARY:
The aim of this study is to promote the inclusive and plural representation of reproductive processes in Spanish fiction, in order to generate knowledge, emotional well-being and improve the quality of life of people in similar situations. The question to be answered is

Will a handbook of good practices used in the training of scriptwriters and audiovisual creators, based on the testimonies of people experiencing reproductive processes and developed with the collaboration of experts (gynaecologists, midwives -ACL-, audiovisuals -Dones Visuals- and scriptwriters -Guionistes Associats-) promote the inclusive and updated representation of reproductive processes?

Focus groups with people involved in reproductive processes and in-depth interviews with professionals involved in these processes will be carried out. A manual of good practices will then be developed in collaboration with audiovisual experts and scriptwriters.

DETAILED DESCRIPTION:
Introduction: Since the 1970s, representations of women in fiction have been the subject of interdisciplinary analysis to understand how cultural narratives perpetuate, challenge or transform patriarchal discourses.

Researchers such as Friedan, Faludi and Macdonald have shown how the media reproduce myths of femininity that reinforce gender inequalities. According to De Lauretis, gender is constructed through representation, while Ricoeur stresses that cultural narratives shape individual identities by linking personal histories with collective imaginaries.

In the area of motherhood, researchers such as Douglas and Michaels, Feasey and Kaplan have shown how the media reinforces conservative ideals such as 'new momism' and simplifies biological processes such as pregnancy and breastfeeding, while personal testimonies reveal tensions between cultural expectations and lived experiences, highlighting the need for more inclusive and diverse narratives.

Aim: The project analyzes the representation of reproductive processes-such as menstruation, pregnancy, abortion, and menopause-in contemporary Spanish audiovisual fiction, assessing how these narratives reflect or challenge socio-cultural structures and reconfigure traditional imaginaries.

Through an intersectional and interdisciplinary approach, the research team aims to understand how different audiences, particularly those related to reproductive health, perceive these narratives. The study will include an analysis of fiction, the perceptions of users and professionals, and collaboration with organizations such as the Catalan Association of Midwives (ACL) and audiovisual experts to co-produce a good practice guide that promotes inclusive, ethical, and patriarchy-free representations.

Material and method: The study will follow a sequential transformative mixed method design (DITRAS), with qualitative predominance and participatory action research, divided into three phases. In the first phase, a quantitative approach will be used with a descriptive cross-sectional study, based on a systematic search of film databases, digital platforms and on-demand television. In the second phase, users' and professionals' perceptions of reproductive health processes will be explored through focus groups and interviews. In the third phase, participatory action research will be applied to co-create a manual of good practices to be implemented in undergraduate and postgraduate training in communication and journalism.

Discussion: To our knowledge, this is the first study to analyze the representation of reproductive processes in Spanish fiction. According to Goffman, the way messages are framed in the media influences the audience's perception of problems and their solutions, leading to psychological, social, and political repercussions.

Through strategically designed narratives, the media has the power to shape attitudes and drive social change, as highlighted by the WHO in its guidelines for addressing sensitive issues such as suicide. Previous studies on the portrayal of childbirth suggest that fiction has distorted the perception of care quality, overrepresented white, heterosexual, non-disabled couples, and depicted women as passive participants in the process.

The findings of this study have the potential to enhance the representation of reproductive processes in the media, fostering a more inclusive and accurate perspective that could shape public perceptions and contribute to the development of more equitable policies.

ELIGIBILITY:
Inclusion Criteria Users:

* Participated in the group health education program at the primary sexual and reproductive health care centers (ASSIR), attended at least 3 sessions.
* Signed the informed consent form.

Exclusion Criteria Users:

- Language barrier (Spanish/Catalan) that limits their ability to have a relaxed conversation.

Inclusion Criteria Health Professionals:

* Employed by the Institut Català de la Salut, specifically within the obstetrics and gynecology team at the Hospital Universitari Arnau de Vilanova (HUAV) or primary health care (ASSIR)
* Signed the informed consent form.

Exclusion Criteria Health Professionals:

- No exclusion criteria were applied.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Use audiovisual works that promote diverse narratives about reproductive processes as case studies in undergraduate and master's programs for future audiovisual professionals | From the implementation of the manual of good practices in university communication and audiovisual studies to 5 years later.
  Implement the use of a best practices manual for students of Audiovisual Communication, Journalism and Screenwriting, to enhance their critical ability to recognize more inclusive narratives in terms of race, class, gender, culture, religion, socioeconomic background, and access to reproductive rights.

SECONDARY OUTCOMES:
Creation of a database of fictional works on reproductive processes in Spain | In the 14 months prior to enrolling to participate.
  To create a database of Spanish fictional works on reproductive processes from the last decade, following a search strategy designed by the research team. To analyze the fiction depicted (keyword, type, author, year, depicted reproductive process, ideology, medicalization, stereotypes, and platform -VOD or free-to-air TV-) using a customized tool for this study.
Profile and perceptions of users and professionals from focus group scripts or semi-structured interviews on the representation of reproductive processes in contemporary Spanish fiction. | An average of 6 months from the registration of participants (users and healthcare professionals) to the completion of the analysis of the interview / focus group.
  A questionnaire will collect sociodemographic data such as age, sex/gender, country of birth, and occupation. Reproductive characteristics such as previous pregnancies, abortions, perinatal losses, live births, obstetric complications, and prior health education will also be gathered. Additionally, users' health education programs and professionals' characteristics (discipline, experience, level of care, and occupation) will be recorded.
  Based on the semi-structured script, users' perceptions of the reproductive process, its differences from real experience, and consequences, including the invisibility of certain processes, will be collected. Discrepancies in care practices and their impact on expectations, along with proposals for improvement, will be analyzed. Professionals' views on fictional representations of sexual-reproductive health, their roles, stereotypes, interprofessional relationships, and impact on the population will also be examined, with suggestions for improvement.
Manual of best practices and recommendations for audiovisual presentations of reproductive processes, based on data collected through focus groups and in-depth interviews with users and professionals. | From the registration of participants in the Participatory Action Intervention Working Group to the implementation of the tool in university communication and audiovisual studies, an average 6 months.
  The co-production of a manual of best practices for audiovisual representations of reproductive processes will be based on the analysis of user and professional discourses, with the participation of sexual and reproductive health experts (gynecologist and Associació Catalana de Llevadores) and communication professionals (Dones Visuals and Guionistes Associats de Catalunya). This manual, aimed at scriptwriters, audiovisual creators and students, will provide recommendations for the accurate representation of reproductive processes, ensuring visibility without gender stereotypes, respecting current health protocols and taking into account the social context.

CONTACTS AND LOCATIONS:
Overall Officials: Mariona Visa Barbosa, PhD, Principal Investigator — Universitat de Lleida; Margarida Carnicé Mur, PhD, Principal Investigator — Universitat de Lleida
Locations (1):
- Facultat d'Infermeria i Fisioteràpia, Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No
The individual data collected in this study contain sensitive personal information. Despite anonymization measures, sharing could compromise participants' privacy and confidentiality. Additionally, the informed consent specifies that the data will be used solely for this study and not shared with third parties. Therefore, individual data sets will not be shared to ensure security and adherence to ethical research principles.

REFERENCES:
- [Background] Acosta Artiles FJ, Rodriguez Rodriguez-Caro CJ, Cejas Mendez MR. [Reporting on Suicide. WHO recommendations for the Media.]. Rev Esp Salud Publica. 2017 Oct 24;91:e201710040. Spanish. PMID 29064462
- [Background] HAYS, Sharon. (1998). The cultural contradictions of motherhood. Yale University press
- [Background] KAPLAN, E. Ann. (2013). Motherhood and representation: The mother in popular culture and melodrama. Routledge.
- [Background] FEASEY, Rebecca. (2016). Mothers on mothers: maternal readings of popular television. Peter Lang
- [Background] FEASEY, Rebecca. (2012). From happy homemaker to desperate housewives: motherhood and popular television. London: Anthem Press.
- [Background] DOUGLAS, Susan y MICHAELS, Meredith. (2004). The Mommy Myth: The Mass Media and the Rise of the New Momism. The Free Press.
- [Background] MACDONALD, Myra (1995) Representing women myths of femininity in the popular media. Hodder Arnold
- [Background] FALUDI, Susan. (1991). Backlash: The undeclared war against women. London: Chatto & Windus
- [Background] Friedan B. The problem that has no name. The Feminine Mystique 1963. Am J Public Health. 2010 Sep;100(9):1582-4. doi: 10.2105/ajph.100.9.1582. No abstract available. PMID 20705962